CLINICAL TRIAL: NCT05705349
Title: A Phase 3, Randomized, Active-Controlled, Double-Blind Clinical Study to Evaluate the Antiretroviral Activity, Safety, and Tolerability of Doravirine/Islatravir (DOR/ISL 100 mg/0.25 mg) Once-Daily in HIV-1 Infected Treatment-Naïve Participants
Brief Title: DOR/ISL in HIV-1 Antiretroviral Treatment-naïve Participants (MK-8591A-053)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 8591A-053; 2022-502099-22-00 (Registry Identifier: EU CT); jRCT2031220720 (Registry Identifier: jRCT); U1111-1283-2516 (Registry Identifier: UTN)
Record Dates: First submitted 2023-01-20; First posted 2023-01-30 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: HIV-1 Infection

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- DOR/ISL (Experimental): Participants take DOR/ISL and placebo to BIC/FTC/TAF once daily (qd) for 144 weeks.
  Interventions: Drug: DOR/ISL; Drug: Placebo to BIC/FTC/TAF
- BIC/FTC/TAF (Active Comparator): Participants take BIC/FTC/TAF and placebo to DOR/ISL qd for 144 weeks.
  Interventions: Drug: BIC/FTC/TAF; Drug: Placebo to DOR/ISL

INTERVENTIONS:
Drug: DOR/ISL — Fixed dose combination tablet containing DOR/ISL 100 mg/0.25 mg taken by mouth.
  Other Names: MK-8591A
  Arms: DOR/ISL
Drug: BIC/FTC/TAF — Fixed dose combination tablet containing BIC/FTC/TAF 50 mg/200 mg/25 mg taken by mouth.
  Arms: BIC/FTC/TAF
Drug: Placebo to DOR/ISL — Placebo tablet matched to DOR/ISL tablet taken by mouth.
  Arms: BIC/FTC/TAF
Drug: Placebo to BIC/FTC/TAF — Placebo tablet matched to BIC/FTC/TAF tablet taken by mouth.
  Arms: DOR/ISL

SUMMARY:
This is a randomized, active-controlled, double-blind clinical study designed to evaluate the antiretroviral activity, safety, and tolerability of doravirine/islatravir (DOR/ISL [MK-8591A]) in treatment-naïve participants with human immunodeficiency virus type 1 (HIV-1) infection. It is hypothesized that DOR/ISL is non-inferior to bictegravir/emtricitabine/tenofovir alafenamide (BIC/FTC/TAF) as assessed by the percentage of participants with HIV-1 ribonucleic acid (RNA) <50 copies/mL at Week 48.

ELIGIBILITY:
Inclusion Criteria:

* Is HIV-1 positive with plasma HIV-1 RNA ≥500 copies/mL at screening
* Is naïve to antiretroviral therapy (ART) defined as having received no prior therapy with any antiretroviral agent following a diagnosis of HIV-1 infection
* If female, is not a participant of childbearing potential (POCBP); or if a POCBP, is not pregnant or breastfeeding, and is willing to use an acceptable contraceptive method or abstain from heterosexual intercourse for study duration

Exclusion Criteria:

* Has HIV-2 infection
* Has hypersensitivity or other contraindication to any of the components of the study interventions as determined by the investigator
* Has a diagnosis of an active AIDS-defining opportunistic infection within 30 days prior to screening
* Has active hepatitis B infection (defined as hepatitis B surface antigen [HBsAg]-positive or HBV deoxyribonucleic acid [DNA]-positive).
* Has chronic hepatitis C virus (HCV) infection (detectable HCV ribonucleic acid [RNA]) and lab values are consistent with cirrhosis
* Has a history of malignancy ≤5 years prior to providing documented informed consent except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or cutaneous Kaposi's sarcoma
* Has a history or current evidence of any condition (including active tuberculosis infection), therapy, laboratory abnormality, or other circumstance (including drug or alcohol use or dependence) that might, in the opinion of the investigator, confound the results of the study or interfere with the participant's participation for the full duration of the study, such that it is not in the best interest of the participant to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 537 (Actual)
Dates: Start 2023-03-08 (Actual); Primary Completion 2025-10-13 (Actual); Study Completion 2029-08-05 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with human immunodeficiency virus type 1 (HIV-1) ribonucleic acid (RNA) <50 copies/mL at Week 48 | Week 48
  Plasma HIV-1 RNA quantification will be performed at the central laboratory using a polymerase chain reaction (PCR) assay with a lower limit of detection of <50 copies/mL.
Percentage of participants experiencing ≥1 adverse event (AE) through Week 48 | Up to 48 weeks
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Percentage of participants discontinuing from study treatment due to an AE through Week 48 | Up to 48 weeks
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.

SECONDARY OUTCOMES:
Percentage of participants with HIV-1 RNA <50 copies/mL at Week 96 | Week 96
  Plasma HIV-1 RNA quantification will be performed at the central laboratory using a PCR assay with a lower limit of detection of <50 copies/mL.
Percentage of participants with HIV-1 RNA <50 copies/mL at Week 144 | Week 144
  Plasma HIV-1 RNA quantification will be performed at the central laboratory using a PCR assay with a lower limit of detection of <50 copies/mL.
Percentage of participants with HIV-1 RNA <200 copies/mL at Week 48 | Week 48
  Plasma HIV-1 RNA quantification will be performed at the central laboratory using a PCR assay with a lower limit of detection of <50 copies/mL.
Percentage of participants with HIV-1 RNA <200 copies/mL at Week 96 | Week 96
  Plasma HIV-1 RNA quantification will be performed at the central laboratory using a PCR assay with a lower limit of detection of <50 copies/mL.
Percentage of participants with HIV-1 RNA <200 copies/mL at Week 144 | Week 144
  Plasma HIV-1 RNA quantification will be performed at the central laboratory using a PCR assay with a lower limit of detection of <50 copies/mL.
Change from baseline in cluster of differentiation 4+ (CD4+) T-cells at Week 48 | Baseline (Day 1) and Week 48
  CD4+ T-cells are quantified with a T and B lymphocyte and natural killer cell (TBNK) panel.
Change from baseline in CD4+ T-cells at Week 96 | Baseline (Day 1) and Week 96
  CD4+ T-cells are quantified with a TBNK panel.
Change from baseline in CD4+ T-cells at Week 144 | Baseline (Day 1) and Week 144
  CD4+ T-cells are quantified with a TBNK panel.
Incidence of viral drug resistance | Up to 96 weeks
  Plasma samples will be collected for genotypic and phenotypic HIV-1 viral drug resistance testing and used to assess resistance-associated substitutions and viral susceptibility as applicable during the study.
Change from baseline in body weight at Week 48 | Baseline (Day 1) and Week 48
  Body weight will be collected throughout the study.
Change from baseline in body weight at Week 96 | Baseline (Day 1) and Week 96
  Body weight will be collected throughout the study.
Change from baseline in body weight at Week 144 | Baseline (Day 1) and Week 144
  Body weight will be collected throughout the study.
Percentage of participants experiencing ≥1 AE through Week 144 | Up to 144 weeks
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Percentage of participants discontinuing from study treatment due to an AE through Week 144 | Up to 144 weeks
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (131):
- United States (38):
  - Pueblo Family Physicians ( Site 5674), Phoenix, Arizona
  - Pacific Oaks Medical Group ( Site 5681), Beverly Hills, California
  - Ruane Clinical Research Group, Inc ( Site 5658), Los Angeles, California
  - Vivent Health ( Site 5694), Denver, Colorado
  - Washington Health Institute ( Site 5689), Washington D.C., District of Columbia
  - Midway Immunology and Research Center ( Site 5657), Ft. Pierce, Florida
  - AHF The Kinder Medical Group ( Site 5672), Miami, Florida
  - AHF South Beach ( Site 5663), Miami Beach, Florida
  - Orlando Immunology Center ( Site 5654), Orlando, Florida
  - CAN Community Health - Sarasota ( Site 5668), Sarasota, Florida
  - Triple O Research Institute, P.A ( Site 5666), West Palm Beach, Florida
  - Emory University and Grady Health System-Medicine ( Site 5690), Atlanta, Georgia
  - Emory University Hospital Midtown Infectious Disease Clinic ( Site 5673), Atlanta, Georgia
  - Atlanta I.D. Group ( Site 5680), Atlanta, Georgia
  - Metro Infectious Diseases Consultants L.L.C. ( Site 5653), Decatur, Georgia
  - Mercer University, Department of Internal Medicine ( Site 5655), Macon, Georgia
  - Rush University Medical Center-Infectious Disease ( Site 5671), Chicago, Illinois
  - University of Illinois at Chicago-Project WISH ( Site 5685), Chicago, Illinois
  - Howard Brown Health Center-Clinical Research ( Site 5665), Chicago, Illinois
  - Be Well Medical Center ( Site 5650), Berkley, Michigan
  - Henry Ford Hospital ( Site 5667), Detroit, Michigan
  - KC CARE Health Center-Clinical Trials ( Site 5670), Kansas City, Missouri
  - Jubilee Clinical Research ( Site 5679), Las Vegas, Nevada
  - Las Vegas Research Center ( Site 5691), Las Vegas, Nevada
  - ID Care ( Site 5676), Hillsborough, New Jersey
  - Saint Michael's Medical Center ( Site 5682), Newark, New Jersey
  - Columbia University Irving Medical Center-Division of Infectious Diseases ( Site 5688), New York, New York
  - Jacobi Medical Center ( Site 5683), The Bronx, New York
  - Atrium Health Infectious Disease Kenilworth - Charlotte ( Site 5675), Charlotte, North Carolina
  - Regional Center for Infectious Diseases ( Site 5687), Greensboro, North Carolina
  - University of Cincinnati Medical Center-Infectious Diseases - Outpatient ( Site 5662), Cincinnati, Ohio
  - Central Texas Clinical Research ( Site 5661), Austin, Texas
  - St Hope Foundation ( Site 5659), Bellaire, Texas
  - Prism Health North Texas, Oak Cliff Health Center ( Site 5660), Dallas, Texas
  - North Texas Infectious Diseases Consultants, P.A ( Site 5651), Dallas, Texas
  - AXCES Research - Texas - El Paso ( Site 5692), El Paso, Texas
  - Texas Centers for Infectious Disease Associates ( Site 5656), Fort Worth, Texas
  - DCOL Center for Clinical Research ( Site 5664), Longview, Texas
- Argentina (5):
  - Fundación Huésped ( Site 5850), CABA, Buenos Aires
  - Instituto de Investigaciones Clínicas Mar del Plata ( Site 5854), Mar del Plata, Buenos Aires
  - Instituto CAICI SRL ( Site 5852), Rosario, Santa Fe Province
  - Fundación IDEAA ( Site 5851), Buenos Aires
  - Instituto Oulton ( Site 5853), Córdoba
- Canada (5):
  - Hamilton Health Sciences-Urgent Care Centre ( Site 5750), Hamilton, Ontario
  - Toronto General Hospital ( Site 5753), Toronto, Ontario
  - Clinique Medicale lActuel ( Site 5752), Montreal, Quebec
  - McGill University Health Centre ( Site 5751), Montreal, Quebec
  - Regina General Hospital ( Site 5754), Regina, Saskatchewan
- Chile (6):
  - Clinica Universidad Catolica del Maule ( Site 5954), Talca, Maule Region
  - Biomedica Research Group-Infectology ( Site 5951), Santiago, Region M. de Santiago
  - Espacio Eme ( Site 5952), Santiago, Region M. de Santiago
  - Centro de Investigacion Clinicadela Universidad Catolica ( Site 5953), Santiago, Region M. de Santiago
  - Universidad de Chile - Hospital Clínico Universidad de Chile-Inmunologia Alergia y VIH ( Site 5950), Santiago, Region M. de Santiago
  - Hospital hernan henriquez aravena de temuco-Unidad de Investigación Clínica ( Site 5955), Temuco, Región de la Araucanía
- Colombia (5):
  - Ciensalud Ips S A S ( Site 6050), Barranquilla, Atlántico
  - Clinica de la Costa S.A.S. ( Site 6055), Barranquilla, Atlántico
  - Hospital Universitario San Ignacio-Infectious ( Site 6053), Bogotá, Bogota D.C.
  - Clinica Colsanitas S.A, Sede Clínica Universitaria Colombia ( Site 6051), Bogotá, Bogota D.C.
  - Fundación Valle del Lili ( Site 6052), Cali, Valle del Cauca Department
- Instituto Dermatológico y Cirugía de Piel "Dr. Huberto Bogaert Díaz" ( Site 8250), Santo Domingo de Guzman, Santo Domingo Province, Dominican Republic
- France (7):
  - Centre Hospitalier Universitaire de Nice - Hôpital l'Archet ( Site 6153), Nice, Alpes-Maritimes
  - Tourcoing Hospital ( Site 6150), Tourcoing, Nord
  - Hôpital Bichat - Claude-Bernard ( Site 6162), Paris
  - Hôpital Saint Antoine ( Site 6158), Paris
  - Hôpital Avicenne ( Site 6160), Bobigny, Île-de-France Region
  - Hôpital Saint-Louis ( Site 6159), Paris, Île-de-France Region
  - Pitie Salpetriere University Hospital ( Site 6156), Paris, Île-de-France Region
- Germany (5):
  - Klinikum der Ludwig-Maximilians-Universitaet Muenchen-Medizinische Klinik und Poliklinik IV, Sektio, München, Bavaria
  - Universitaetsklinikum Freiburg ( Site 6256), Freiburg, Brandenburg
  - Universitätsklinikum Bonn-Immunologie ( Site 6250), Bonn, North Rhine-Westphalia
  - ICH Study Center GmbH & Co. KG ( Site 6259), Hamburg
  - Universitaetsklinikum Hamburg-Eppendorf-Infektiologie ( Site 6260), Hamburg
- Guatemala (3):
  - CLINIPHARM ( Site 8352), Guatemala City
  - Clínica Médica Especializada en Pediatría e Infectología Pediátrica - Dr. Mario Melgar ( Site 8350), Guatemala City
  - CELAN,S.A ( Site 8351), Guatemala City
- Israel (4):
  - Rambam Health Care Campus-Institute of Allergy, Clinical Immunology, ( Site 6751), Haifa
  - Hadassah Medical Center-Infecious Disease ( Site 6752), Jerusalem
  - Sheba Medical Center-HIV unit ( Site 6753), Ramat Gan
  - Sourasky Medical Center ( Site 6754), Tel Aviv
- Japan (4):
  - National Hospital Organization Nagoya Medical Center ( Site 6953), Nagoya, Aichi-ken
  - Tokyo Medical University Hospital ( Site 6954), Shinjuku-ku, Tokyo
  - Center Hospital of the National Center for Global Health and Medicine ( Site 6951), Shinjyuku-ku, Tokyo
  - National Hospital Organization Osaka National Hospital ( Site 6952), Osaka
- Kenya (3):
  - CCR KEMRI (Center for Clinical Research) ( Site 8652), Nairobi, Nairobi City
  - PHRD KEMRI (Partners in Health Research & Development) ( Site 8651), Nairobi, Nairobi City
  - KEMRI-CMR-RCTP ( Site 8650), Kisumu
- Malaysia (7):
  - Hospital Sultanah Bahiyah ( Site 7776), Alor Star, Kedah
  - University Malaya Medical Centre-Clinical Investigation Centre (CIC) ( Site 7777), Lembah Pantai, Kuala Lumpur
  - Hospital Pulau Pinang ( Site 7779), George Town, Pulau Pinang
  - Sarawak General Hospital ( Site 7772), Kuching, Sarawak
  - Hospital Selayang ( Site 7770), Batu Caves, Selangor
  - Hospital Sungai Buloh ( Site 7778), Sungai Buloh, Selangor
  - Hospital Kuala Lumpur ( Site 7773), Kuala Lumpur
- Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran ( Site 7251), Mexico City, Mexico City, Mexico
- Puerto Rico (3):
  - Ponce Medical School Foundation Inc. ( Site 7452), Ponce
  - Clinical Research Puerto Rico ( Site 7450), San Juan
  - HOPE Clinical Research ( Site 7451), San Juan
- South Africa (11):
  - Josha Research ( Site 6652), Bloemfontein, Free State
  - Perinatal HIV Research Unit (PHRU)-Adult Treatment and Research ( Site 6654), Johannesburg, Gauteng
  - Helen Joseph Hospital-Clinical HIV Research Unit ( Site 6661), Johannesburg, Gauteng
  - Ezintsha-Clinical Research Site ( Site 6656), Johannesburg, Gauteng
  - Wentworth Hospital ( Site 6653), Durban, KwaZulu-Natal
  - Qhakaza Mbokodo Research Clinic ( Site 6659), Ladysmith, KwaZulu-Natal
  - Human Sciences Research Council-Centre for Community Based Research ( Site 6664), Pietermaritzburg, KwaZulu-Natal
  - Madibeng Centre for Research ( Site 6660), Brits, North West
  - Family Clinical Research Unit (Fam-Cru)-Adult Infectious Diseases ( Site 6657), Cape Town, Western Cape
  - Desmond Tutu Health Foundation ( Site 6651), Cape Town, Western Cape
  - Be Part Yoluntu Centre ( Site 6650), Paarl, Western Cape
- Spain (11):
  - Hospital General Universitario de Elche-Infectius Disease ( Site 6358), Elche, Alicante
  - Hospital Germans Trias i Pujol-Fundació Lluita contra la Sida ( Site 6351), Badalona, Barcelona
  - HOSPITAL CLÍNIC DE BARCELONA-Infection Day Hospital ( Site 6350), Barcelona, Catalonia
  - Hospital Universitari de Bellvitge ( Site 6360), L'Hospitalet de Llobregat,Barcelona, Catalonia
  - HOSPITAL GENERAL UNIVERSITARIO GREGORIO MARAÑON-Unidad de Enfermedades Infecciosas ( Site 6353), Madrid, Madrid, Comunidad de
  - Hospital Universitario Ramón y Cajal-ENFERMEDADES INFECCIOSAS ( Site 6361), Madrid, Madrid, Comunidad de
  - Hospital Universitari Vall d'Hebron-Infectious Diseases: HIV unit ( Site 6352), Barcelona
  - Hospital Universitario Fundación Jiménez Díaz-Internal Medicine. Infectious disease ( Site 6357), Madrid
  - Hospital Universitario 12 de Octubre ( Site 6355), Madrid
  - Hospital Universitario La Paz ( Site 6354), Madrid
  - Hospital Universitario Virgen de la Victoria ( Site 6359), Málaga
- Switzerland (2):
  - University Hospital Basel-Infectiology ( Site 8151), Basel, Canton of Basel-City
  - Hôpitaux Universitaires de Genève (HUG)-Infectious Disease Department ( Site 8150), Geneva, Canton of Geneva
- Thailand (3):
  - HIV Netherlands Australia Thailand Research Collaboration ( Site 7851), Bangkok, Bangkok
  - Faculty of Medicine Siriraj Hospital-Preventive and social ( Site 7850), Bangkok, Bangkok
  - Research Institute for Health Sciences-Research Institute for Health Sciences Building 1 ( Site 7852, Chiang Mai
- Turkey (Türkiye) (2):
  - Hacettepe Universite Hastaneleri ( Site 7650), Altindağ, Ankara
  - Ankara Bilkent Şehir Hastanesi-Infectious Disease and Clinical Microbiology ( Site 7659), Ankara
- United Kingdom (5):
  - Southmead Hospital ( Site 7952), Bristol, Bristol, City of
  - Royal London Hospital ( Site 7951), London, England
  - The Hathersage Centre ( Site 7953), Manchester, England
  - King's College Hospital ( Site 7950), London, London, City of
  - The Mortimer Market Centre for Sexual Health and HIV Research ( Site 7954), London, London, City of

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26120&tenant=MT_MSD_9011